CLINICAL TRIAL: NCT03446170
Title: Examining the Impact of Cigarette Package Warnings and Packaging Regulations Among Young Adult Smokers
Brief Title: Effect of Cigarette Pack Warnings and Packaging Among Young Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Darren Mays, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2014-1031
Record Dates: First submitted 2018-02-12; First posted 2018-02-26 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Tobacco Use
Keywords: Young adults; Cigarette smoking; Warning labels
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: The experimental design is a 2 (graphic warning message framing: gain versus loss) by 2 (cigarette packaging: standardized, plain or branded) factorial design. An unexposed control group is also included.
Masking Description: The study tests the effects of graphic cigarette warning labels and packaging regulations, therefore it is unmasked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Loss-framed, branded (Experimental): Participants assigned to this arm use cigarette packs with loss-framed graphic warnings communicating the risks of smoking on branded packages.
  Interventions: Behavioral: Graphic cigarette warning labels, plain packaging
- Loss-framed, plain (Experimental): Participants assigned to this arm use cigarette packs with loss-framed graphic warnings communicating the risks of smoking on plain or standardized packages.
  Interventions: Behavioral: Graphic cigarette warning labels, plain packaging
- Gain-framed, branded (Experimental): Participants assigned to this arm use cigarette packs with gain-framed graphic warnings communicating the benefits of quitting smoking on branded packages.
  Interventions: Behavioral: Graphic cigarette warning labels, plain packaging
- Gain-framed, plain (Experimental): Participants assigned to this arm use cigarette packs with gain-framed graphic warnings communicating the benefits of quitting smoking on plain or standardized packages.
  Interventions: Behavioral: Graphic cigarette warning labels, plain packaging
- Control (No Intervention): Participants assigned to this arm use their regular cigarette packs and complete study measures only.

INTERVENTIONS:
Behavioral: Graphic cigarette warning labels, plain packaging — This study tests the effects of graphic cigarette warning labels that include pictures and text, and plain or standardized packaging
  Arms: Gain-framed, branded; Gain-framed, plain; Loss-framed, branded; Loss-framed, plain

SUMMARY:
The objective of this study is to examine whether cigarette packaging regulations including graphic health warning labels on cigarette packs and requiring plain, unbranded packaging reduce the appeal of cigarettes and prompt young adult smokers to quit.

DETAILED DESCRIPTION:
The study includes young adult smokers ages 18 to 30. Eligible participants are young adults ages 18 to 30 years inclusive who report smoking at least 100 lifetime cigarettes and now smoking on all or some days. Participants must also reside in the metro Washington, DC area. The first portion of the study is a within-subjects experiment simulating point of sale cigarette purchase behaviors based on 2 packaging features: (1) graphic warning messages framed to emphasize either the health benefits of quitting (i.e., gain framed) or the health risks of smoking (i.e., loss-framed) and (2) industry branded or plain (i.e., standardized unbranded) packaging. In the second portion of the study, the same participants take part in a prospective experiment to determine the impact of graphic cigarette warning message framing (gain versus loss) and packaging (branded versus plain) on motivation to quit and smoking behavior. Participants are randomized to use 1 of 4 experimentally adapted cigarette packs in place of their regular packs for 4 weeks, or to a control condition which will continue to use their regular packs. All participants complete baseline and follow-up assessments and respond to daily mobile phone text message prompts on their personal mobile phones during the 4 week exposure period. Participants complete follow-up assessments capturing motivation to quit, smoking behavior, and quit attempts at the conclusion of the 4 week exposure period and 1- and 3-months later.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 30 years
* Smoke at least 100 cigarettes in their lifetime
* Now smoke cigarettes on all or some days
* Reside in the Washington, DC metro area
* Willing to send and receive text messages on a personal mobile phone

Exclusion Criteria:

* No additional exclusion criteria

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Cigarette purchase appeal | Baseline
  The effects of graphic cigarette warnings and plain packaging on cigarette purchase appeal will be measured using data collected from a within-subjects experiment at baseline. Participants are randomly assigned to compare each pair of packs from the experimental conditions versus a standard branded control pack. For each pair, cigarette purchase appeal is measured with 5 valid questions assessing: 1) Which pack would you be most likely to buy? 2) Which pack is the most appealing? 3) Which pack attracts your attention? 4) Which pack contains cigarettes that are the most harmful to your health? 5) Which pack makes you think about the health risks of smoking?
Motivation to quit smoking | At the conclusion of the 4 week exposure
  Motivation to quit smoking is measured using a valid scale comprised of 4 questions. Participants report how likely it is they will quit smoking completely, reduce the number of cigarettes they smoke, and talk to a friend, family member, or spouse/partner about quitting smoking. Participants respond using options for definitely will not, probably will not, probably will, or definitely will for each question.

SECONDARY OUTCOMES:
Cigarette smoking behavior | At the conclusion of the 4 week exposure, and at 1- and 3-months post-exposure
  Cigarettes smoked per day is measured using a single valid question assessing about how many cigarettes participants smoked each day, on average.
Smoking quit attempts | At the conclusion of the 4 week exposure, and at 1- and 3-months post-exposure
  Attempts to quit smoking is measured using a single valid item asking participants how many times they stopped smoking for 1 day or longer because they were trying to quit.
Motivation to quit cigarette smoking. | At 1-month and 3-months post-exposure
  Motivation to quit smoking is measured using a valid scale comprised of 4 questions. Participants report how likely it is they will quit smoking completely, reduce the number of cigarettes they smoke, and talk to a friend, family member, or spouse/partner about quitting smoking. Participants respond using options for definitely will not, probably will not, probably will, or definitely will for each question.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mays, PhD, MPH, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will consider requests to share de-identified individual participant data by request and according to our study protocol and institutional data sharing policy.

REFERENCES:
- [Background] Johnson AC, Luta G, Tercyak KP, Niaura RS, Mays D. Effects of pictorial warning label message framing and standardized packaging on cigarette packaging appeal among young adult smokers. Addict Behav. 2021 Sep;120:106951. doi: 10.1016/j.addbeh.2021.106951. Epub 2021 Apr 13. PMID 33895661
- [Background] Johnson AC, Turner MM, Simmens SJ, Evans WD, Strasser AA, Mays D. Mediational Effects on Motivation to Quit Smoking After Exposure to a Cigarette Pictorial Warning Label Among Young Adults. Ann Behav Med. 2022 Jul 12;56(7):737-748. doi: 10.1093/abm/kaab073. PMID 34415010
- [Background] Johnson AC, Simmens SJ, Turner MM, Evans WD, Strasser AA, Mays D. Longitudinal effects of cigarette pictorial warning labels among young adults. J Behav Med. 2022 Feb;45(1):124-132. doi: 10.1007/s10865-021-00258-2. Epub 2021 Sep 23. PMID 34554369